CLINICAL TRIAL: NCT05842265
Title: The Effect of Self Acupressure Application on Pain, Fatigue and Sleep Quality in Multiple Myeloma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/ 15- 43
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Self Acupressure; Sleep; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): Self acupressure
  Interventions: Other: Self acupressure
- Control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Other: Self acupressure — patients will do self acupressure
  Arms: Experimental:

SUMMARY:
Multiple Myeloma occurs with damaging bone lesion, hypercalcemia, anemia and renal failure as a result of secretion of monoclonal protein in serum and/or urea and accumulation of plasma cells. The most common symptoms at the time of diagnosis are; fatigue, insomnia, bone pain and recurrent infections. In multiple myeloma patients, pain, fatigue and sleep problems are conditions that significantly affect the daily life activities of the individual and require planned nursing interventions for the solution. In this challenging process, a holistic approach should be adopted while planning the care practices of the patients, and non-pharmacological practices should be planned, which will enable the patient to perform the activities of daily life with minimum energy and maximum function. Acupressure, one of the non-pharmacological applications, is a complementary medicine method that ensures the proper functioning of the energy channels by applying pressure to the points on the energy-carrying meridians (these points are the same as acupuncture points) with fingers, palms or wrist bands without using needles, unlike acupuncture. In the literature, it is stated that acupressure is a pain-relieving, relaxing analgesic and immune system-strengthening supportive method rather than its therapeutic effect, and it relieves insomnia and fatigue and relieves the person. In addition, within the scope of the harmonization model; By teaching acupressure to patients by nurses, patients can be actively involved in their own symptom management. Therefore, this study was planned to evaluate the effect of self-acupressure applied to patients with multiple myeloma on pain, fatigue and sleep quality.

The research will be conducted as a randomized, experimental study with a pretest-posttest control group. The sample of the study will consist of 52 Multiple Myeloma patients, 26 experimental and 26 control groups, who met the research criteria and accepted the study, between August 2022 and January 2023, in Hematology Clinic and Polyclinic of Fırat University Hospital. Patients in the experimental group will be asked to perform self-acupressure by showing and teaching the LI4, HT 7, ST36 and SP6 acupressure points by the researcher. Depending on the preparation and compression time on these 4 points, the patients will be asked to perform a total of 16 sessions for 4 weeks, for a total of 18 minutes, 2 days a week in the morning and afternoon. The 1st measurement will be obtained by applying the Patient Information Form, Visual Analog Scale "Pitssburg Sleep Quality Index (PUKI)" and Piper Fatigue Scale" to the patients in the experimental group at the pre-test stage before the application. After 4 weeks, the Pitssburg Sleep Quality Index (PUKI) and The second measurement will be obtained by applying the "Piper Fatigue Scale" again. No application will be made to the patients in the control group. In the pre-test phase, the 1st measurement will be obtained by applying only the Patient Information Form, Visual Analog Scale, Pitssburg Sleep Quality Index (PUKI) and Piper Fatigue Scale. After 4 weeks, in the post-test phase, the second measurement will be obtained by re-applying the other forms except the Patient Information Form. The data will be analyzed using the SPSS 23 program. Shapiro Wilk test, t test, Mann-Whitney U test, Wilcoxon test and Chi-square analysis will be used in the analysis of the data.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a disease characterized by monoclonal neoplastic proliferation of immunoglobulin-producing plasma cells (1). Plasma cells proliferate in the bone marrow and cause extensive damage to the skeletal system, often with osteolytic lesions, osteopenia, and/or pathological fractures. Anemia is a malignant disease characterized by the presence of monoclonal protein in serum and urine, hypercalcemia, and renal failure (1).

Multiple Myeloma is a disease of advanced age. The mean age at diagnosis of the patients is 66. It constitutes 1% of all malignancies and 10% of hematological malignancies (2). Although its etiology is not known exactly, it is thought that obesity, smoking, diet, radiation, immune system and environmental factors may be responsible (3).

Plasma cells develop from B lymphocytes (4). Bone marrow microenvironment is important in the development of Multiple Myeloma. Advanced stage memory B cell/plasmablast, which has provided the isotypic change of Immune globulin (Ig) in the germinal center, is the premyeloma cell in which the oncogenic effect begins. It then settles in the bone marrow a second oncogenic effect occurs in the cell (5). Multiple Myeloma is a disease with a wide clinical spectrum. Symptoms and signs related to anemia, radicular back and low back pain due to pathological vertebral fractures, bone pain due to osteolytic lesions, pathological fractures, peripheral polyneuropathy, renal failure, hypercalcemia, hyperviscosity syndrome, thrombosis and bleeding tendency, infection can be seen in patients (6). It is evaluated whether the patient is a candidate for autologous stem cell transplantation (OKHN) in the treatment of Multiple Myeloma. In young patients with MM, high-dose chemotherapy and OKHN are applied as standard treatment. OKHN increases cure rates, prolongs progression-free and overall survival (7). The application of a triple combination containing bortezomib is used as a standard in induction therapy in international myeloma centers (7,8). Depending on their physical condition and specific complications, patients who are not suitable for stem cell transplantation are treated differently.treatment options are available. Treatment options including bortezomib in patients with renal insufficiency and lenalidomide in patients with neuropathy can be given (9). There is usually no cure in Multiple Myeloma, the majority of patients receive second-line and other-line treatments.

ELIGIBILITY:
Inclusion Criteria:

Having a scale score of >5 on the Piper Fatigue Scale Having a score of >5 on the Pittsburgh Sleep Quality Scale Pain severity is 5 points or higher according to the Visual Analog Scale

Exclusion criteria; Using acupressure and similar integrative treatment methods, Having a verbal communication disability (hearing and speaking), Having a diagnosed psychiatric disorder,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Pitssburg Sleep Quality Index | 4 week
  It was developed by Buysse et al. (1989) (34). The scale is a safe and consistent questionnaire that evaluates the amount of sleep, sleep quality, presence and severity of sleep disorders in individuals in the last month. It was adapted into Turkish by Ağargün et al. (1996) (35). There are seven components in PUKI. These components are subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), sleep medication use (component 6) and daytime dysfunction. (component 7). The evaluation score of each item is between 0-3. The total score obtained varies between 0-21. The higher the score, the worse the sleep quality.
Piper Fatigue Scale | 4 week
  The Piper Fatigue Scale was developed in 1987 by Piper et al. It was developed by.The Turkish validity and reliability study of the scale was conducted by Can in 2001 (37). The scale evaluates the individual's subjective perception of fatigue in four sub-dimensions. These; behavior/violence sub-dimension evaluating the effect and severity of fatigue on activities of daily living (ADLs (6 items; 2-7); affect sub-dimension, which includes the emotional meaning attributed to fatigue (5 items; 8-12); it is the sensory sub-dimension (5 items; 13-17) that reflects the mental, physical and emotional symptoms of fatigue, and the cognitive/spiritual sub-dimension that reflects the effect of fatigue on cognitive functions and mental state (6 items; 18-23). As a result of the average score; 0 points are interpreted as no fatigue, 1-3 points as mild fatigue, 4-6 points as moderate fatigue, 7-10 points as severe fatigue.
Visual Analog Scale | 4 week
  Patients are asked to show the intensity of pain on a 10 cm long vertical or horizontal line during activity or rest. It has numbered shapes ranging from 1-10. The line has 0 at the beginning and 10 at the end. 10 means unbearable pain, 0 means no pain. The VAS scale is frequently used in the evaluation of pain severity. While the patient marks the pain he/she has felt on this line, each point marked is measured in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan B.TURAN, Principal Investigator — Elazığ /Merkez/Turkey/23000
Locations (1):
- Gülcan B Turan, Elâzığ, Merkez, Turkey (Türkiye)